CLINICAL TRIAL: NCT00653354
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Dose Assessment Of The Analgesic Efficacy Of The Dosing Regimen Of Valdecoxib Compared To Placebo Patients In Pain Following Bunionectomy
Brief Title: Analgesic Efficacy Of Valdecoxib In Patients Following Bunion Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VALA-0513-149; A3471086
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Pain, Post-surgical
Keywords: hallux valgus
MeSH Terms: conditions — Pain, Postoperative; Hallux Valgus | interventions — valdecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Active Comparator)
  Interventions: Drug: valdecoxib
- Arm 2 (Active Comparator)
  Interventions: Drug: valdecoxib/placebo
- Arm 3 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: valdecoxib — valdecoxib 40 mg tablet by mouth within 6 hours of surgery followed by valdecoxib 20 mg tablet by mouth 1 to 12 hours after the first dose
  Arms: Arm 1
Drug: valdecoxib/placebo — valdecoxib 40 mg tablet by mouth within 6 hours of surgery followed by placebo 1 to 12 hours after the first dose
  Arms: Arm 2
Drug: placebo — placebo within 6 hours of surgery followed by placebo 1 to 12 hours after the first dose
  Arms: Arm 3

SUMMARY:
To assess the analgesic efficacy and general safety of 2 dosing regimens of valdecoxib compared to placebo on the first post-operative day in patients with moderate or severe pain following bunionectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent an uncomplicated primary unilateral first metatarsal bunionectomy surgery (with or without ipsilateral hammer toe repair) requiring open manipulation of bone with periosteal elevation under regional anesthesia (Mayo block)
* Patients had a Baseline pain intensity of moderate or severe on a categorical scale and ≥45 mm on a VAS

Exclusion Criteria:

* Patients who were scheduled to undergo other surgical procedures that would be expected to produce a greater degree of surgical trauma than the orthopedic procedure alone
* Patients treated with patient controlled analgesia (PCA) subsequent to the end of anesthesia
* Patients treated with long-acting local anesthetics or local anesthetics coadministered with epinephrine injected into the index joint space
* Patients expected to require analgesics or other agents other than study medication during the 8 hours preceding administration of study medication through the end of the treatment period, that could confound assessment of the analgesic response, specifically excluded were tricyclic antidepressants, tranquilizers, neuroleptics, neuroleptic antiemetics, cyclooxygenase-2 inhibitors, nonsteroidal antiinflammatory drugs, and corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2002-12; Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Summed Pain Intensity Difference (categorical) through 24 hours (SPID 24) | Day 1
Total Pain Relief through 24 hours (TOTPAR 24) | Day 1
Patient's Global Evaluation of Study Medication | Day 1

SECONDARY OUTCOMES:
time between doses of study medication | Day 1
Time-specific Pain Intensity Difference (PID) (categorical) | 0, 2, 4, 6, 8, 10, 12, 16, and 24 hours
time-specific pain relief | 2, 4, 6, 8, 10, 12, 16, and 24 hours
time-specific PID (VAS) | 0, 2, 4, 6, 8, 10, 12, 16, and 24 hours
Summed Pain Intensity (SPID)24 (VAS) | 0, 2, 4, 6, 8, 10, 12, 16, and 24 hours
time to rescue medication | 2, 4, 6, 8, 10, 12, 16, and 24 hours
percent of patients who took rescue medication | Day 1
Patient's Satisfaction Questionnaire | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- United States (13):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tempe, Arizona
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Chula Vista, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Santa Ana, California
  - Pfizer Investigational Site, Tustin, California
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Altoona, Pennsylvania
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Johnson City, Tennessee
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah